CLINICAL TRIAL: NCT01931839
Title: A Phase 3, Rollover Study to Evaluate the Safety and Efficacy of Long-term Treatment With Lumacaftor in Combination With Ivacaftor in Subjects Aged 12 Years and Older With Cystic Fibrosis, Homozygous or Heterozygous for the F508del-CFTR Mutation
Brief Title: A Phase 3 Rollover Study of Lumacaftor in Combination With Ivacaftor in Subjects 12 Years and Older With Cystic Fibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VX12-809-105
Record Dates: First submitted 2013-08-26; First posted 2013-08-29 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Cystic Fibrosis, Homozygous or Heterozygous for the F508del-CFTR Mutation
MeSH Terms: conditions — Cystic Fibrosis | interventions — lumacaftor; ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Arm 1 Part A: LUM 600 mg qd/ IVA 250 mg q12h (Experimental): Participants who received lumacaftor (LUM, VX-809) 600 milligram (mg) plus ivacaftor (IVA, VX-770) 250 mg fixed-dose combination (FDC) tablet orally in the morning and IVA 250 mg film-coated tablet orally in the evening, in the previous study VX12-809-103 or VX12-809-104, and will receive the same treatment in this study VX12-809-105 up to Week 96.
  Interventions: Drug: Lumacaftor Plus Ivacaftor Combination; Drug: Ivacaftor
- Arm 2 Part A: Placebo - LUM 600 mg qd/ IVA 250 mg q12h (Experimental): Participants who received placebo matched to LUM and IVA tablet in the previous study VX12-809-103 or VX12-809-104, and will receive LUM 600 mg plus IVA 250 mg FDC tablet orally in the morning and IVA 250 mg film-coated tablet orally in the evening in this study VX12-809-105 up to Week 96.
  Interventions: Drug: Lumacaftor Plus Ivacaftor Combination; Drug: Ivacaftor
- Arm 3 Part A: LUM 400 mg q12h/ IVA 250 mg q12h (Experimental): Participants who received LUM 400 mg plus IVA 250 mg FDC tablet orally in the morning and evening in the previous study VX12-809-103 or VX12-809-104, and will receive the same treatment in this study VX12-809-105 up to Week 96.
  Interventions: Drug: Lumacaftor Plus Ivacaftor Combination
- Arm 4 Part A: Placebo - LUM 400 mg q12h/ IVA 250 mg q12h (Experimental): Participants who received placebo matched to LUM and IVA tablet in the previous study VX12-809-103 or VX12-809-104, and will receive LUM 400 mg plus IVA 250 mg FDC tablet orally in the morning and evening in this study VX12-809-105 up to Week 96.
  Interventions: Drug: Lumacaftor Plus Ivacaftor Combination
- Arm 5 Part A: Observational Cohort (No Intervention): Participants who received either LUM 600 mg plus IVA 250 mg FDC tablet orally in the morning and IVA 250 mg film-coated tablet orally in the evening OR LUM 400 mg plus IVA 250 mg FDC tablet orally in the morning and evening OR placebo matched to LUM and IVA in the morning and evening, in the previous study VX12-809-103 or VX12-809-104, and will be observed (will not receive study drug) in this study VX12-809-105 for up to 2 years.
- Arm 6 Part B: LUM 400 mg q12h/ IVA 250 mg q12h (Experimental): Participants who received LUM 400 mg plus IVA 250 mg FDC tablet orally in the morning and evening in Cohort 4 of the previous study VX09-809-102, and will receive the same treatment in this study VX12-809-105 up to Week 96.
  Interventions: Drug: Lumacaftor Plus Ivacaftor Combination
- Arm 7 Part B: Placebo - LUM 400 mg q12h/ IVA 250 mg q12h (Experimental): Participants who received placebo matched to LUM and IVA tablet in Cohort 4 of the previous study VX09-809-102, and will receive LUM 400 mg plus IVA 250 mg FDC tablet orally in the morning and evening in this study VX12-809-105 up to Week 96.
  Interventions: Drug: Lumacaftor Plus Ivacaftor Combination

INTERVENTIONS:
Drug: Lumacaftor Plus Ivacaftor Combination — Fixed dose combination tablet, oral use
  Arms: Arm 1 Part A: LUM 600 mg qd/ IVA 250 mg q12h; Arm 2 Part A: Placebo - LUM 600 mg qd/ IVA 250 mg q12h; Arm 3 Part A: LUM 400 mg q12h/ IVA 250 mg q12h; Arm 4 Part A: Placebo - LUM 400 mg q12h/ IVA 250 mg q12h; Arm 6 Part B: LUM 400 mg q12h/ IVA 250 mg q12h; Arm 7 Part B: Placebo - LUM 400 mg q12h/ IVA 250 mg q12h
Drug: Ivacaftor — Film-coated tablet, oral use
  Arms: Arm 1 Part A: LUM 600 mg qd/ IVA 250 mg q12h; Arm 2 Part A: Placebo - LUM 600 mg qd/ IVA 250 mg q12h

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of long-term treatment with lumacaftor in combination with ivacaftor in people 12 years and older with Cystic Fibrosis.

DETAILED DESCRIPTION:
This is a Phase 3, parallel group, multicenter, rollover study in participants with CF who are homozygous or heterozygous for the F508del CFTR mutation and who previously participated in Study 103 (Study VX12-809-103, NCT01807923), Study 104 (Study VX12-809-104, NCT01807949), or Cohort 4 of Study 102 (Study VX09-809-102, NCT01225211).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF), and where appropriate, signed assent form.
* Participants entering the Part A Treatment Cohort: Completed 24 weeks of study drug treatment in Study 103 or Study 104 and elect to enroll in Part A treatment cohort.
* Participants entering the Part B Treatment Cohort: Completed 56 days of study drug treatment in Cohort 4 of Study 102 and elect to enroll in Part B treatment cohort.
* Participants entering the Part A Observational Cohort: Completed 24 weeks of study drug treatment in Study 103 or Study 104, but do not elect to enroll in the Part A Treatment Cohort or do not qualify to enroll in Part A treatment cohort.
* Willing to remain on a stable CF medication regimen through the end of study (Part A and Part B Treatment Cohorts only).

Exclusion Criteria:

* Any comorbidity or laboratory abnormality that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the participant (e.g., cirrhosis with portal hypertension).
* Pregnant and nursing females. Females of childbearing potential must have a negative pregnancy test at the Day 1 Visit.
* History of drug intolerance in the prior study that would pose an additional risk to the participant in the opinion of investigator or Vertex.
* History of poor compliance with study drug and/or procedures in the previous study as deemed by the investigator.
* Participation in an investigational drug trial (including studies investigating lumacaftor and/or ivacaftor, or studies requiring blood collections with or without administration of study drug)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1164 (Actual)
Dates: Start 2013-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (166):
- United States (91):
  - Birmingham, Alabama
  - Anchorage, Alaska
  - Tucson, Arizona
  - Little Rock, Arkansas
  - La Jolla, California
  - Loma Linda, California
  - Longbeach, California
  - Los Angeles, California
  - Madera, California
  - Oakland, California
  - Palo Alto, California
  - Sacramento, California
  - Aurora, Colorado
  - Denver, Colorado
  - Hartford, Connecticut
  - New Haven, Connecticut
  - Altamonte Springs, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - Park Ridge, Illinois
  - Peoria, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Kansas City, Kansas
  - Lexington, Kentucky
  - New Orleans, Louisiana
  - South Portland, Maine
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Grand Rapids, Michigan
  - Minneapolis, Minnesota
  - Jackson, Mississippi
  - Kansas City, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Bedford, New Hampshire
  - Lebanon, New Hampshire
  - Long Branch, New Jersey
  - Morristown, New Jersey
  - New Brunswick, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Buffalo, New York
  - Lake Success, New York
  - New York, New York
  - Rochester, New York
  - Syracuse, New York
  - Valhalla, New York
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charelston, South Carolina
  - Sioux Falls, South Dakota
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Tyler, Texas
  - Salt Lake City, Utah
  - Colchester, Vermont
  - Charlottesville, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Spokane, Washington
  - Morgantown, West Virginia
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Australia (8):
  - New Lambton Heights, New South Wales
  - Westmead, New South Wales
  - Adelaide, Queensland
  - Chermside, Queensland
  - Herston, Queensland
  - South Brisbane, Queensland
  - Nedlands
  - Subiaco
- Austria (2):
  - Innsbruck
  - Wels
- Belgium (4):
  - Brussels
  - Ghent
  - Leuven
  - Liège
- Canada (7):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Halifax, Nova Scotia
  - Ottowa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Czechia (3):
  - Brno
  - Plzeň - Bory
  - Prague
- Copenhagen, Denmark
- France (11):
  - Strasbourg, Bas Rhin
  - Marseille, Bouches-du-Rhone
  - Toulouse, Haute Garonne
  - Montpellier, Herault
  - Lille, Nord
  - Bron, Rhone
  - Bordeaux
  - Paris
  - Pierre-Bénite
  - Rhone
  - Roscoff
- Germany (15):
  - Munich, Bavaria
  - München, Bayem
  - München, Muenchen
  - Berlin
  - Bochum
  - Cologne
  - Erlangen
  - Essen
  - Frankfurt
  - Giessen
  - Hanover
  - Jena
  - Leipzig
  - Tübingen
  - Würzburg
- Dublin, Ireland
- Italy (6):
  - Ancona
  - Florence
  - Genova
  - Milan
  - Roma
  - Verona
- Netherlands (4):
  - Amsterdam
  - Nijmegen
  - Rotterdam
  - The Hague
- Spain (2):
  - Barcelona
  - Valencia
- Sweden (2):
  - Gothenburg
  - Stockholm
- United Kingdom (9):
  - Exeter, Devon
  - Belfast
  - Birmingham
  - Bristol
  - Leeds
  - London
  - Newcastle
  - Nottingham
  - Southampton

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662
- [Derived] Konstan MW, McKone EF, Moss RB, Marigowda G, Tian S, Waltz D, Huang X, Lubarsky B, Rubin J, Millar SJ, Pasta DJ, Mayer-Hamblett N, Goss CH, Morgan W, Sawicki GS. Assessment of safety and efficacy of long-term treatment with combination lumacaftor and ivacaftor therapy in patients with cystic fibrosis homozygous for the F508del-CFTR mutation (PROGRESS): a phase 3, extension study. Lancet Respir Med. 2017 Feb;5(2):107-118. doi: 10.1016/S2213-2600(16)30427-1. Epub 2016 Dec 21. PMID 28011037

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study conducted in 2 parts: A & B. Part A consisted of Treatment Cohorts & Observational Cohort, which enrolled participants from Study VX12-809-103 (Study 103, NCT01807923) & Study VX12-809-104 (Study 104, NCT01807949). Part B consisted of Treatment Cohorts which enrolled participants from Cohort 4 of Study VX09-809-102 (Study 102, NCT01225211).
Pre-assignment Details: Of 1164 participants enrolled, 1163 were dosed and included in this study.
Groups:
- Arm 1 Part A: LUM 600 mg qd/ IVA 250 mg q12h: Participants who received lumacaftor (LUM, VX-809) 600 milligram (mg) plus ivacaftor (IVA, VX-770) 250 mg fixed-dose combination (FDC) tablet orally in the morning and IVA 250 mg film-coated tablet orally in the evening, in the previous study VX12-809-103 or VX12-809-104, received the same treatment in this study VX12-809-105 up to Week 96.
- Arm 2 Part A: Placebo - LUM 600 mg qd/ IVA 250 mg q12h: Participants who received placebo matched to LUM and IVA tablet in the previous study VX12-809-103 or VX12-809-104, received LUM 600 mg plus IVA 250 mg FDC tablet orally in the morning and IVA 250 mg film-coated tablet orally in the evening in this study VX12-809-105 up to Week 96.
- Arm 3 Part A: LUM 400 mg q12h/ IVA 250 mg q12h: Participants who received LUM 400 mg plus IVA 250 mg FDC tablet orally in the morning and evening in the previous study VX12-809-103 or VX12-809-104, received the same treatment in this study VX12-809-105 up to Week 96.
- Arm 4 Part A: Placebo - LUM 400 mg q12h/ IVA 250 mg q12h: Participants who received placebo matched to LUM and IVA tablet in the previous study VX12-809-103 or VX12-809-104, received LUM 400 mg plus IVA 250 mg FDC tablet orally in the morning and evening in this study VX12-809-105 up to Week 96.
- Arm 5 Part A: Observational Cohort: Participants who received either LUM 600 mg plus IVA 250 mg FDC tablet orally in the morning and IVA 250 mg film-coated tablet orally in the evening OR LUM 400 mg plus IVA 250 mg FDC tablet orally in the morning and evening OR placebo matched to LUM and IVA in the morning and evening, in the previous study VX12-809-103 or VX12-809-104, were observed (did not receive study drug) in this study VX12-809-105 for up to 2 years.
- Arm 6 Part B: LUM 400 mg q12h/ IVA 250 mg q12h: Participants who received LUM 400 mg plus IVA 250 mg FDC tablet orally in the morning and evening in Cohort 4 of the previous study VX09-809-102, received the same treatment in this study VX12-809-105 up to Week 96.
- Arm 7 Part B: Placebo - LUM 400 mg q12h/ IVA 250 mg q12h: Participants who received placebo matched to LUM and IVA tablet in Cohort 4 of the previous study VX09-809-102, received LUM 400 mg plus IVA 250 mg FDC tablet orally in the morning and evening in this study VX12-809-105 up to Week 96.
Period: Overall Study
Arm/Group | Arm 1 Part A: LUM 600 mg qd/ IVA 250 mg q12h | Arm 2 Part A: Placebo - LUM 600 mg qd/ IVA 250 mg q12h | Arm 3 Part A: LUM 400 mg q12h/ IVA 250 mg q12h | Arm 4 Part A: Placebo - LUM 400 mg q12h/ IVA 250 mg q12h | Arm 5 Part A: Observational Cohort | Arm 6 Part B: LUM 400 mg q12h/ IVA 250 mg q12h | Arm 7 Part B: Placebo - LUM 400 mg q12h/ IVA 250 mg q12h
Started | 335 | 178 | 340 | 176 | 19 | 55 | 60
Full Analysis Set (As Randomized) | 334 | 179 | 340 | 176 | 19 | 55 | 60
Safety Analysis Set (As Dosed) | 335 | 178 | 340 | 176 | 19 | 55 | 60
Completed | 294 | 152 | 301 | 162 | 18 | 50 | 56
Not Completed | 41 | 26 | 39 | 14 | 1 | 5 | 4
Not completed — Death | 0 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Withdrawal of consent | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 9 | 4 | 1 | 3 | 0 | 0 | 1
Not completed — Withdrawal of consent (not due to AE) | 11 | 8 | 13 | 3 | 0 | 2 | 2
Not completed — Other non-compliance | 15 | 9 | 12 | 3 | 0 | 3 | 0
Not completed — Lost to Follow-up | 1 | 2 | 4 | 5 | 0 | 0 | 0
Not completed — Other | 4 | 2 | 6 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set (study 105) included all participants who were exposed to any amount of study drug.
Groups:
- q12h Arm 2 Part A: Placebo - LUM 600 mg qd/ IVA 250 mg q12h: Participants who received placebo matched to LUM and IVA tablet in the previous study VX12-809-103 or VX12-809-104, received LUM 600 mg plus IVA 250 mg FDC tablet orally in the morning and IVA 250 mg film-coated tablet orally in the evening in this study VX12-809-105 up to Week 96.
- Total: Total of all reporting groups
Arm/Group | Arm 1 Part A: LUM 600 mg qd/ IVA 250 mg q12h | q12h Arm 2 Part A: Placebo - LUM 600 mg qd/ IVA 250 mg q12h | Arm 3 Part A: LUM 400 mg q12h/ IVA 250 mg q12h | Arm 4 Part A: Placebo - LUM 400 mg q12h/ IVA 250 mg q12h | Arm 5 Part A: Observational Cohort | Arm 6 Part B: LUM 400 mg q12h/ IVA 250 mg q12h | Arm 7 Part B: Placebo - LUM 400 mg q12h/ IVA 250 mg q12h | Total
Number analyzed (Participants) | 335 | 178 | 340 | 176 | 19 | 55 | 60 | 1163
Age, Customized [Count of Participants; unit: Participants]
  12 years to less than 18 years | 93 | 47 | 94 | 47 | 2 | 0 | 0 | 283
  Greater than or equal to 18 years | 242 | 131 | 246 | 129 | 17 | 55 | 60 | 880
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166 | 89 | 164 | 86 | 12 | 25 | 31 | 573
  Male | 169 | 89 | 176 | 90 | 7 | 30 | 29 | 590

OUTCOME MEASURES:

1. Primary Outcome: Part A Treatment Cohort: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: as any untoward medical occurrence in a participant during the study; the event does not necessarily have a causal relationship with the treatment. This includes any newly occurring event or previous condition that has increased in severity or frequency after informed consent form is signed. AE includes serious as well as non-serious AEs. SAE (subset of AE): medical event or condition, which falls into any of the following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, In-patient hospitalization/prolongation of hospitalization, persistent/significant disability or incapacity, congenital anomaly/birth defect, important medical event. Any AE that increased in severity or newly developed at or after initial dosing of study drug was considered treatment-emergent.
Time Frame: Day 1 up to Week 105 (Study 105)
Population: Safety Set (study 105) included all participants in Treatment Cohort Part A who were exposed to any amount of study drug.
Measure: Number; unit: participants
Groups:
- Arm 1: Part A - LUM 600 mg qd/ IVA 250 mg q12h: Participants who received LUM 600 mg plus IVA 250 mg FDC tablet orally in the morning and IVA 250 mg film-coated tablet orally in the evening, in the previous study VX12-809-103 (NCT01807923) or VX12-809-104 (NCT01807949), received the same treatment in this study VX12-809-105 (NCT01931839) up to Week 96.
- Arm 2: Part A - Placebo- LUM 600 mg qd/ IVA 250 mg q12h: Participants who received placebo matched to LUM and IVA tablet in the previous study VX12-809-103 (NCT01807923) or VX12-809-104 (NCT01807949), received LUM 600 mg plus IVA 250 mg FDC tablet orally in the morning and IVA 250 mg film-coated tablet orally in the evening in this study VX12-809-105 (NCT01931839) up to Week 96.
- Arm 3: Part A - LUM 400 mg q12h/ IVA 250 mg q12h: Participants who received LUM 400 mg plus IVA 250 mg FDC tablet orally in the morning and evening in the previous study VX12-809-103 (NCT01807923) or VX12-809-104 (NCT01807949), received the same treatment in this study VX12-809-105 (NCT01931839) up to Week 96.
- Arm 4: Part A - Placebo- LUM 400 mg q12h/ IVA 250 mg q12h: Participants who received placebo matched to LUM and IVA tablet in the previous study VX12-809-103 (NCT01807923) or VX12-809-104 (NCT01807949), received LUM 400 mg plus IVA 250 mg FDC tablet orally in the morning and evening in this study VX12-809-105 (NCT01931839) up to Week 96.
Arm/Group | Arm 1: Part A - LUM 600 mg qd/ IVA 250 mg q12h | Arm 2: Part A - Placebo- LUM 600 mg qd/ IVA 250 mg q12h | Arm 3: Part A - LUM 400 mg q12h/ IVA 250 mg q12h | Arm 4: Part A - Placebo- LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 335 | 178 | 340 | 176
participants
  Participants with any AEs | 331 | 177 | 333 | 176
  Participants with SAEs | 156 | 77 | 143 | 89

2. Primary Outcome: Part B Treatment Cohort: Number of Participants With Treatment-Emergent AEs and SAEs
Description: as for outcome 1
Time Frame: Day 1 up to Week 105 (Study 105)
Population: Safety Set (study 105) included all participants in the Treatment Cohort Part B who were exposed to any amount of study drug.
Measure: Number; unit: participants
Groups:
- Arm 6: Part B LUM 400 mg q12h/ IVA 250 mg q12h: Participants who received LUM 400 mg plus IVA 250 mg FDC tablet orally in the morning and evening in Cohort 4 of the previous study VX09-809-102 (NCT01225211), received the same treatment in this VX12-809-105 (NCT01931839) up to Week 96.
- Arm 7: Part B Placebo- LUM 400 mg q12h/ IVA 250 mg q12h: Participants who received placebo matched to LUM and IVA tablet in Cohort 4 of the previous study VX09-809-102 (NCT01225211), received LUM 400 mg plus IVA 250 mg FDC tablet orally in the morning and evening in this study VX12-809-105 (NCT01931839) up to Week 96.
Arm/Group | Arm 6: Part B LUM 400 mg q12h/ IVA 250 mg q12h | Arm 7: Part B Placebo- LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 55 | 60
participants
  Participants with AEs | 52 | 57
  Participants with SAEs | 18 | 21

3. Secondary Outcome: Part A Treatment Cohort: Absolute Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) At Day 15, Week 8, 16, 24, 36, 48, 60 and 72
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Hankinson and Wang standards were used to calculate percent predicted FEV1 (for age, gender, race, and height). The Hankinson standard was used for male participants 18 years and older and female participants 16 years and older. The Wang standard was used for male participants aged 12 to 17 years and for female participants aged 12 to 15 years. Analysis was performed using baseline of the previous study VX12-809-103 (NCT01807923) and Study VX12-809-104 (NCT01807949) for Arm 1 and 3. Analysis was performed using baseline of the current study VX12-809-105 (NCT01931839) for Arm 2 and 4.
Time Frame: Baseline (Study 103/104/105); Day 15, Week 8, 16, 24, 36, 48, 60 , 72 (Study 105)
Population: Full Analysis Set (FAS) study 105 (NCT01931839) included all participants randomized in the Part A Treatment Cohort and dosed. Here, 'Number of participants analyzed' = those participants who were evaluable for this endpoint and 'Number Analyzed' = those participants who were evaluable at the specified time points for each arm, respectively.
Measure: Least Squares Mean (Standard Error); unit: percent predicted of FEV1
Arm/Group | Arm 1: Part A - LUM 600 mg qd/ IVA 250 mg q12h | Arm 2: Part A - Placebo- LUM 600 mg qd/ IVA 250 mg q12h | Arm 3: Part A - LUM 400 mg q12h/ IVA 250 mg q12h | Arm 4: Part A - Placebo- LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 319 | 173 | 317 | 165
percent predicted of FEV1
  Absolute Change at Day 15 | 3 (0.5) | 2.8 (0.6) | 2.8 (0.5) | 3 (0.6)
  Absolute Change at Week 8: number analyzed (Participants) | 309 | 164 | 316 | 165
  Absolute Change at Week 8 | 3.1 (0.5) | 2.8 (0.6) | 3.4 (0.5) | 4.2 (0.6)
  Absolute Change at Week 16: number analyzed (Participants) | 307 | 166 | 313 | 160
  Absolute Change at Week 16 | 2.6 (0.5) | 2.7 (0.6) | 2.5 (0.5) | 3.6 (0.7)
  Absolute Change at Week 24: number analyzed (Participants) | 291 | 158 | 295 | 154
  Absolute Change at Week 24 | 2.9 (0.5) | 2.4 (0.6) | 2.7 (0.5) | 3.4 (0.7)
  Absolute Change at Week 36: number analyzed (Participants) | 292 | 155 | 294 | 150
  Absolute Change at Week 36 | 2.7 (0.5) | 2.2 (0.7) | 1.9 (0.5) | 3.1 (0.7)
  Absolute Change at Week 48: number analyzed (Participants) | 279 | 153 | 286 | 143
  Absolute Change at Week 48 | 1.5 (0.5) | 1.8 (0.7) | 1.4 (0.5) | 2.1 (0.7)
  Absolute Change at Week 60: number analyzed (Participants) | 276 | 146 | 282 | 140
  Absolute Change at Week 60 | 1.7 (0.5) | 2.1 (0.7) | 1.6 (0.5) | 1.4 (0.7)
  Absolute Change at Week 72: number analyzed (Participants) | 275 | 146 | 273 | 134
  Absolute Change at Week 72 | 1.2 (0.5) | 1.9 (0.7) | 0.5 (0.5) | 1.5 (0.7)

4. Secondary Outcome: Part B Treatment Cohort: Absolute Change From Baseline in Percent Predicted FEV1 at Day 15, Week 8, 16, 24, 36, 48, 60 and 72
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Hankinson and Wang standards were used to calculate percent predicted FEV1 (for age, gender, race, and height). The Hankinson standard was used for male participants 18 years and older and female participants 16 years and older. The Wang standard was used for male participants aged 12 to 17 years and for female participants aged 12 to 15 years. Analysis was performed using baseline of Cohort 4 of previous study VX09-809-102 (NCT01225211) for Arm 6 and 7.
Time Frame: Baseline (Study 102), Day 15, Week 8, 16, 24, 36, 48, 60 , 72 (Study 105)
Population: FAS (study 105) included all participants randomized in the Part B Treatment Cohort and dosed. Here, 'Number of participants analyzed' = those participants who were evaluable for this endpoint and 'Number Analyzed' = those participants who were evaluable at the specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: percent predicted of FEV1
Arm/Group | Arm 6: Part B LUM 400 mg q12h/ IVA 250 mg q12h | Arm 7: Part B Placebo- LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 52 | 57
percent predicted of FEV1
  Absolute Change at Day 15 | -2 (8) | -3.4 (6.6)
  Absolute Change at Week 8: number analyzed (Participants) | 49 | 55
  Absolute Change at Week 8 | -3.9 (7.4) | -1.8 (6.4)
  Absolute Change at Week 16: number analyzed (Participants) | 50 | 52
  Absolute Change at Week 16 | -3.1 (9) | -2.8 (6.8)
  Absolute Change at Week 24: number analyzed (Participants) | 36 | 36
  Absolute Change at Week 24 | -2.9 (7.7) | -2.5 (7.3)
  Absolute Change at Week 36: number analyzed (Participants) | 20 | 19
  Absolute Change at Week 36 | -3.2 (7.9) | -2.3 (7.9)
  Absolute Change at Week 48: number analyzed (Participants) | 15 | 17
  Absolute Change at Week 48 | -5.4 (11.2) | -2 (6)
  Absolute Change at Week 60: number analyzed (Participants) | 12 | 16
  Absolute Change at Week 60 | -1.8 (10.1) | -1.9 (8.2)
  Absolute Change at Week 72: number analyzed (Participants) | 11 | 15
  Absolute Change at Week 72 | -2.8 (9.2) | -7.8 (8.3)

5. Secondary Outcome: Part A Treatment Cohort: Relative Change From Baseline in Percent Predicted FEV1 at Day 15, Week 8, 16, 24, 36, 48, 60 and 72
Description: as for outcome 3
Time Frame: Baseline (Study 103/104/105), Day 15, Week 8, 16, 24, 36, 48, 60 , 72 (Study 105)
Population: FAS study 105 (NCT01931839) included all participants randomized in the Part A Treatment Cohort and dosed. Here, 'Number of participants analyzed' = those participants who were evaluable for this endpoint and 'Number Analyzed' = those participants who were evaluable at the specified time points for each arm, respectively.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Arm 1: Part A - LUM 600 mg qd/ IVA 250 mg q12h | Arm 2: Part A - Placebo- LUM 600 mg qd/ IVA 250 mg q12h | Arm 3: Part A - LUM 400 mg q12h/ IVA 250 mg q12h | Arm 4: Part A - Placebo- LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 319 | 173 | 317 | 165
percent change
  Relative Change at Day 15 | 5.3 (0.9) | 5.1 (1.2) | 5.3 (0.9) | 4.8 (1.2)
  Relative Change at Week 8: number analyzed (Participants) | 309 | 164 | 316 | 165
  Relative Change at Week 8 | 5.6 (0.9) | 5.6 (1.2) | 6.2 (0.9) | 7.1 (1.2)
  Relative Change at Week 16: number analyzed (Participants) | 307 | 166 | 313 | 160
  Relative Change at Week 16 | 4.9 (0.9) | 5.4 (1.2) | 4.8 (0.9) | 6.5 (1.2)
  Relative Change at Week 24: number analyzed (Participants) | 291 | 158 | 295 | 154
  Relative Change at Week 24 | 5.1 (0.9) | 4.9 (1.2) | 5 (0.9) | 6.1 (1.2)
  Relative Change at Week 36: number analyzed (Participants) | 292 | 155 | 294 | 150
  Relative Change at Week 36 | 4.7 (0.9) | 4 (1.2) | 3.6 (0.9) | 5.5 (1.2)
  Relative Change at Week 48: number analyzed (Participants) | 279 | 153 | 286 | 143
  Relative Change at Week 48 | 2.7 (0.9) | 3.6 (1.2) | 2.9 (0.9) | 3.6 (1.2)
  Relative Change at Week 60: number analyzed (Participants) | 276 | 146 | 282 | 140
  Relative Change at Week 60 | 2.9 (0.9) | 4.1 (1.2) | 2.7 (0.9) | 3.1 (1.2)
  Relative Change at Week 72: number analyzed (Participants) | 275 | 146 | 273 | 134
  Relative Change at Week 72 | 2.4 (0.9) | 3.8 (1.2) | 1.4 (0.9) | 2.6 (1.2)

6. Secondary Outcome: Part B Treatment Cohort: Relative Change From Baseline in Percent Predicted FEV1 at Day 15, Week 8, 16, 24, 36, 48, 60 and 72
Description: as for outcome 4
Time Frame: Baseline (Study 102), Day 15, Week 8, 16, 24, 36, 48, 60 , 72 (Study 105)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Arm 6: Part B LUM 400 mg q12h/ IVA 250 mg q12h | Arm 7: Part B Placebo- LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 52 | 57
percent change
  Relative Change at Day 15 | -2.2 (13.6) | -5.8 (11.4)
  Relative Change at Week 8: number analyzed (Participants) | 49 | 55
  Relative Change at Week 8 | -5.2 (12.8) | -3.1 (11.4)
  Relative Change at Week 16: number analyzed (Participants) | 50 | 52
  Relative Change at Week 16 | -4.2 (15.8) | -4.9 (11.8)
  Relative Change at Week 24: number analyzed (Participants) | 36 | 36
  Relative Change at Week 24 | -3.4 (13.2) | -4.2 (12.6)
  Relative Change at Week 36: number analyzed (Participants) | 20 | 19
  Relative Change at Week 36 | -4.1 (12.5) | -3.5 (14.2)
  Relative Change at Week 48: number analyzed (Participants) | 15 | 17
  Relative Change at Week 48 | -6.9 (15.9) | -2.8 (10.6)
  Relative Change at Week 60: number analyzed (Participants) | 12 | 16
  Relative Change at Week 60 | -0.7 (16.6) | -2.6 (13.9)
  Relative Change at Week 72: number analyzed (Participants) | 11 | 15
  Relative Change at Week 72 | -3.3 (13.3) | -11.8 (10.7)

7. Secondary Outcome: Part A Treatment Cohort: Absolute Change From Baseline in Body Mass Index (BMI) at Day 15, Week 8, 16, 24, 36, 48, 60 and 72
Description: BMI = (Weight in kilogram [kg]) divided by (Stature in meters [m]) ^2. Analysis was performed using baseline of the previous study VX12-809-103 (NCT01807923) and Study VX12-809-104 (NCT01807949) for Arm 1 and 3. Analysis was performed using baseline of the current study VX12-809-105 (NCT01931839) for Arm 2 and 4.
Time Frame: Baseline (Study 103/104/105), Day 15, Week 8, 16, 24, 36, 48, 60 , 72 (Study 105)
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Kilogram per square meter (kg/m^2)
Arm/Group | Arm 1: Part A - LUM 600 mg qd/ IVA 250 mg q12h | Arm 2: Part A - Placebo- LUM 600 mg qd/ IVA 250 mg q12h | Arm 3: Part A - LUM 400 mg q12h/ IVA 250 mg q12h | Arm 4: Part A - Placebo- LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 329 | 178 | 338 | 175
Kilogram per square meter (kg/m^2)
  Absolute Change at Day 15: number analyzed (Participants) | 328 | 178 | 338 | 175
  Absolute Change at Day 15 | 0.56 (0.06) | 0.06 (0.08) | 0.5 (0.06) | 0.1 (0.08)
  Absolute Change at Week 8: number analyzed (Participants) | 329 | 173 | 331 | 172
  Absolute Change at Week 8 | 0.58 (0.06) | 0.14 (0.08) | 0.55 (0.06) | 0.27 (0.08)
  Absolute Change at Week 16: number analyzed (Participants) | 321 | 173 | 325 | 170
  Absolute Change at Week 16 | 0.58 (0.06) | 0.19 (0.08) | 0.53 (0.06) | 0.35 (0.08)
  Absolute Change at Week 24: number analyzed (Participants) | 312 | 169 | 319 | 165
  Absolute Change at Week 24 | 0.61 (0.06) | 0.22 (0.08) | 0.62 (0.06) | 0.41 (0.08)
  Absolute Change at Week 36: number analyzed (Participants) | 304 | 165 | 315 | 160
  Absolute Change at Week 36 | 0.66 (0.06) | 0.33 (0.08) | 0.72 (0.06) | 0.59 (0.08)
  Absolute Change at Week 48: number analyzed (Participants) | 299 | 162 | 307 | 151
  Absolute Change at Week 48 | 0.63 (0.06) | 0.42 (0.08) | 0.71 (0.06) | 0.62 (0.09)
  Absolute Change at Week 60: number analyzed (Participants) | 296 | 158 | 298 | 147
  Absolute Change at Week 60 | 0.71 (0.06) | 0.54 (0.08) | 0.8 (0.06) | 0.62 (0.09)
  Absolute Change at Week 72: number analyzed (Participants) | 287 | 152 | 289 | 145
  Absolute Change at Week 72 | 0.72 (0.06) | 0.52 (0.08) | 0.69 (0.06) | 0.62 (0.09)

8. Secondary Outcome: Part B Treatment Cohort: Absolute Change From Baseline in BMI at Day 15, Week 8, 16, 24, 36, 48, 60 and 72
Description: BMI = (Weight [in kg]) divided by (Stature [in meters]) ^2. Analysis was performed using baseline of Cohort 4 of previous study VX09-809-102 (NCT01225211) for Arm 6 and 7.
Time Frame: Baseline (Study 102), Day 15, Week 8, 16, 24, 36, 48, 60 , 72 (Study 105)
Population: FAS (study 105) included all participants randomized in the Part B Treatment Cohort and dosed. Here, 'Number Analyzed' = those participants who were evaluable at the specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Arm 6: Part B LUM 400 mg q12h/ IVA 250 mg q12h | Arm 7: Part B Placebo- LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 55 | 60
kg/m^2
  Absolute Change at Day 15 | -0.05 (0.52) | -0.03 (0.69)
  Absolute Change at Week 8: number analyzed (Participants) | 54 | 57
  Absolute Change at Week 8 | -0.01 (0.82) | 0.14 (0.84)
  Absolute Change at Week 16: number analyzed (Participants) | 51 | 53
  Absolute Change at Week 16 | 0.08 (1.02) | 0.2 (1.09)
  Absolute Change at Week 24: number analyzed (Participants) | 39 | 37
  Absolute Change at Week 24 | 0.04 (0.92) | 0.14 (1.08)
  Absolute Change at Week 36: number analyzed (Participants) | 20 | 20
  Absolute Change at Week 36 | 0.07 (0.54) | 0.85 (1.23)
  Absolute Change at Week 48: number analyzed (Participants) | 17 | 17
  Absolute Change at Week 48 | 0.05 (0.64) | 0.81 (1.55)
  Absolute Change at Week 60: number analyzed (Participants) | 12 | 16
  Absolute Change at Week 60 | 0.08 (0.7) | 0.58 (1.23)
  Absolute Change at Week 72: number analyzed (Participants) | 13 | 15
  Absolute Change at Week 72 | 0.08 (0.71) | 0.41 (1.28)

9. Secondary Outcome: Part A Treatment Cohort: Number of Pulmonary Exacerbations Events Per Patient-Year
Description: Pulmonary exacerbation was defined as the treatment with new or changed antibiotic therapy (intravenous, inhaled, or oral) for greater than or equal to 4 sinopulmonary signs/symptoms. The number of events per patient year were reported, where patient years = total number of days on study/336. Analysis includes all events in the Cumulative Study Period for Arm 1 and 3, and all events in the Current Study period (Study 105) for Arm 2 and 4. As per planned analysis, endpoint evaluation included subjects from the parent study VX12-809-103 and VX12-809-104 as well for cumulative study period.
Time Frame: Baseline (Study 103/104) up to Week 100 (Study 105) for Arm 1 and 3 (Cumulative study period); Baseline (Study 105) up to Week 100 (Study 105) for Arm 2 and 4 (current study period)
Population: FAS (Study 103/104) was used for Arm 1 & 3, & included all participants randomized in previous studies & dosed. FAS (Study 105) was used for Arm 2 & 4, & included all participants randomized in Part A Treatment Cohort & dosed in current study 105. 'Number Analyzed'=those participants who were evaluable at specified time points for each arm.
Measure: Number (95% Confidence Interval); unit: events per patient year
Groups:
- Arm 1: Part A - LUM 600 mg qd/ IVA 250 mg q12h: Participants who were randomized to LUM 600 mg plus IVA 250 mg FDC tablet orally in the morning and IVA 250 mg film-coated tablet orally in the evening in the previous study VX12-809-103 (NCT01807923) or VX12-809-104 (NCT01807949).
- Arm 3: Part A - LUM 400 mg q12h/ IVA 250 mg q12h: Participants who were randomized to LUM 400 mg plus IVA 250 mg FDC tablet orally in the morning and evening in the previous study VX12-809-103 (NCT01807923) or VX12-809-104 (NCT01807949).
Arm/Group | Arm 1: Part A - LUM 600 mg qd/ IVA 250 mg q12h | Arm 2: Part A - Placebo- LUM 600 mg qd/ IVA 250 mg q12h | Arm 3: Part A - LUM 400 mg q12h/ IVA 250 mg q12h | Arm 4: Part A - Placebo- LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 368 | 179 | 369 | 176
events per patient year | 0.38 [0.32 to 0.46] | 0.42 [0.33 to 0.54] | 0.32 [0.26 to 0.38] | 0.37 [0.29 to 0.49]

10. Secondary Outcome: Part A Treatment Cohort: Absolute Change From Baseline in Cystic Fibrosis Questionnaire - Revised (CFQ-R) Respiratory Domain Score at Day 15, Week 8, 16, 24, 48 and 72
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms (for example, coughing, congestion, wheezing), the scaled score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life. Analysis was performed using baseline of the previous study VX12-809-103 (NCT01807923) and Study VX12-809-104 (NCT01807949) for Arm 1 and 3. Analysis was performed using baseline of the current study VX12-809-105 (NCT01931839) for Arm 2 and 4.
Time Frame: Baseline (Study 103/104/105), Day 15, Week 8, 16, 24, 48, 72 (Study 105)
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Arm 1: Part A - LUM 600 mg qd/ IVA 250 mg q12h | Arm 2: Part A - Placebo- LUM 600 mg qd/ IVA 250 mg q12h | Arm 3: Part A - LUM 400 mg q12h/ IVA 250 mg q12h | Arm 4: Part A - Placebo- LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 324 | 174 | 325 | 170
units on a scale
  Absolute Change at Day 15 | 5.9 (0.9) | 2.3 (1.2) | 6.2 (0.9) | 3.5 (1.2)
  Absolute Change at Week 8: number analyzed (Participants) | 323 | 164 | 319 | 166
  Absolute Change at Week 8 | 5 (0.9) | 4.1 (1.2) | 5.1 (0.9) | 6.8 (1.2)
  Absolute Change at Week 16: number analyzed (Participants) | 313 | 167 | 312 | 160
  Absolute Change at Week 16 | 4.1 (0.9) | 2.8 (1.2) | 6.4 (0.9) | 7 (1.2)
  Absolute Change at Week 24: number analyzed (Participants) | 305 | 161 | 304 | 155
  Absolute Change at Week 24 | 6 (0.9) | 3.8 (1.2) | 6.1 (0.9) | 4.7 (1.3)
  Absolute Change at Week 48: number analyzed (Participants) | 290 | 152 | 290 | 140
  Absolute Change at Week 48 | 2 (0.9) | 3.1 (1.3) | 3.7 (0.9) | 1.5 (1.3)
  Absolute Change at Week 72: number analyzed (Participants) | 265 | 141 | 269 | 135
  Absolute Change at Week 72 | 3.2 (0.9) | 3.3 (1.3) | 5.7 (0.9) | 3.3 (1.3)

11. Secondary Outcome: Part B Treatment Cohort: Absolute Change From Baseline in CFQ-R Respiratory Domain Score at Day 15, Week 8, 16, 24, 48 and 72
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms (for example, coughing, congestion, wheezing), the scaled score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life. Analysis was performed using baseline of Cohort 4 of previous study VX09-809-102 (NCT01225211) for Arm 6 and 7.
Time Frame: Baseline (Study 102 Study), Day 15, Week 8, 16, 24, 48, 72 (Study 105)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 6: Part B LUM 400 mg q12h/ IVA 250 mg q12h | Arm 7: Part B Placebo- LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 55 | 59
units on a scale
  Absolute Change at Day 15 | 3.9 (18) | -4.1 (18.1)
  Absolute Change at Week 8: number analyzed (Participants) | 54 | 57
  Absolute Change at Week 8 | 4.8 (18.6) | 1 (18.2)
  Absolute Change at Week 16: number analyzed (Participants) | 51 | 53
  Absolute Change at Week 16 | 6.2 (17.2) | -0.2 (17)
  Absolute Change at Week 24: number analyzed (Participants) | 39 | 37
  Absolute Change at Week 24 | 6.8 (19.1) | -1.2 (17.9)
  Absolute Change at Week 48: number analyzed (Participants) | 19 | 17
  Absolute Change at Week 48 | 2 (14) | 4.9 (15.6)
  Absolute Change at Week 72: number analyzed (Participants) | 13 | 15
  Absolute Change at Week 72 | 8.5 (21.8) | 2.2 (18.8)

12. Secondary Outcome: Part A Treatment Cohort: Absolute Change From Baseline in BMI Z-score at Day 15, Week 8, 16, 24, 36, 48, 60 and 72
Description: z-score is a statistical measure to evaluate how a single data point compares to a standard. It describes whether a mean was above or below the standard and how unusual the measurement is with range from -infinity to +infinity; 0: same mean, >0: a greater mean, and <0: a lesser mean than the standard. BMI-for-age z-score was calculated by using centers for disease control and prevention (CDC) growth charts for the pediatric population. Analysis was performed using baseline of the previous study VX12-809-103 (NCT01807923) and Study VX12-809-104 (NCT01807949) for Arm 1 and 3. Analysis was performed using baseline of the current study VX12-809-105 (NCT01931839) for Arm 2 and 4.
Time Frame: Baseline (Study 103/104/105), Day 15, Week 8, 16, 24, 36, 48, 60, 72 (Study 105)
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Arm 1: Part A - LUM 600 mg qd/ IVA 250 mg q12h | Arm 2: Part A - Placebo- LUM 600 mg qd/ IVA 250 mg q12h | Arm 3: Part A - LUM 400 mg q12h/ IVA 250 mg q12h | Arm 4: Part A - Placebo- LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 117 | 56 | 109 | 60
z-score
  Absolute Change at Day 15 | 0.16 (0.04) | -0.01 (0.06) | 0.14 (0.04) | -0.02 (0.05)
  Absolute Change at Week 8: number analyzed (Participants) | 114 | 53 | 105 | 60
  Absolute Change at Week 8 | 0.15 (0.04) | 0.04 (0.06) | 0.16 (0.04) | 0.08 (0.05)
  Absolute Change at Week 16: number analyzed (Participants) | 112 | 53 | 101 | 58
  Absolute Change at Week 16 | 0.12 (0.04) | 0.08 (0.06) | 0.15 (0.04) | 0.07 (0.05)
  Absolute Change at Week 24: number analyzed (Participants) | 110 | 49 | 100 | 56
  Absolute Change at Week 24 | 0.14 (0.04) | 0.08 (0.06) | 0.17 (0.04) | 0.1 (0.05)
  Absolute Change at Week 36: number analyzed (Participants) | 100 | 46 | 100 | 52
  Absolute Change at Week 36 | 0.14 (0.04) | 0.13 (0.06) | 0.16 (0.04) | 0.14 (0.05)
  Absolute Change at Week 48: number analyzed (Participants) | 95 | 46 | 97 | 47
  Absolute Change at Week 48 | 0.09 (0.04) | 0.13 (0.06) | 0.11 (0.04) | 0.12 (0.06)
  Absolute Change at Week 60: number analyzed (Participants) | 91 | 45 | 90 | 44
  Absolute Change at Week 60 | 0.11 (0.04) | 0.16 (0.06) | 0.14 (0.04) | 0.13 (0.06)
  Absolute Change at Week 72: number analyzed (Participants) | 85 | 45 | 89 | 42
  Absolute Change at Week 72 | 0.06 (0.04) | 0.12 (0.06) | 0.04 (0.04) | 0.08 (0.06)

13. Secondary Outcome: Part A Treatment Cohort: Absolute Change From Baseline in Body Weight at Day 15, Week 8, 16, 24, 36, 48, 60 and 72
Description: Analysis was performed using baseline of the previous study VX12-809-103 (NCT01807923) and Study VX12-809-104 (NCT01807949) for Arm 1 and 3. Analysis was performed using baseline of the current study VX12-809-105 (NCT01931839) for Arm 2 and 4.
Time Frame: Baseline (Study 103/104/105), Day 15, Week 8, 16, 24, 36, 48, 60, 72 (Study 105)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Arm 1: Part A - LUM 600 mg qd/ IVA 250 mg q12h | Arm 2: Part A - Placebo- LUM 600 mg qd/ IVA 250 mg q12h | Arm 3: Part A - LUM 400 mg q12h/ IVA 250 mg q12h | Arm 4: Part A - Placebo- LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 329 | 178 | 338 | 175
kilograms (kg)
  Absolute Change at Day 15: number analyzed (Participants) | 328 | 178 | 338 | 175
  Absolute Change at Day 15 | 1.7 (2.6) | -0.1 (1.8) | 1.3 (2.9) | 0.1 (1.2)
  Absolute Change at Week 8: number analyzed (Participants) | 329 | 173 | 331 | 172
  Absolute Change at Week 8 | 1.8 (2.9) | 0.2 (2.1) | 1.5 (3.1) | 0.6 (1.9)
  Absolute Change at Week 16: number analyzed (Participants) | 321 | 173 | 325 | 170
  Absolute Change at Week 16 | 1.9 (3.2) | 0.4 (2.6) | 1.6 (3.3) | 1 (2.5)
  Absolute Change at Week 24: number analyzed (Participants) | 312 | 169 | 319 | 165
  Absolute Change at Week 24 | 2.2 (3.5) | 0.6 (2.6) | 2 (3.6) | 1.2 (2.8)
  Absolute Change at Week 36: number analyzed (Participants) | 304 | 165 | 315 | 160
  Absolute Change at Week 36 | 2.3 (3.8) | 1 (3.4) | 2.4 (3.8) | 1.9 (3.4)
  Absolute Change at Week 48: number analyzed (Participants) | 299 | 162 | 307 | 151
  Absolute Change at Week 48 | 2.4 (4.2) | 1.3 (3.7) | 2.5 (4.3) | 2.1 (3.7)
  Absolute Change at Week 60: number analyzed (Participants) | 296 | 158 | 298 | 147
  Absolute Change at Week 60 | 2.7 (4.6) | 1.7 (4.2) | 2.9 (4.6) | 2.2 (4.4)
  Absolute Change at Week 72: number analyzed (Participants) | 287 | 152 | 289 | 145
  Absolute Change at Week 72 | 2.9 (4.9) | 1.7 (4.8) | 2.7 (4.9) | 2.3 (4.7)

14. Secondary Outcome: Part B Treatment Cohort: Absolute Change From Baseline in Body Weight at Day 15, Week 8, 16, 24, 36, 48, 60 and 72
Description: Analysis was performed using baseline of Cohort 4 of previous study VX09-809-102 (NCT01225211) for Arm 6 and 7.
Time Frame: Baseline (Study 102), Day 15, Week 8, 16, 24, 36, 48, 60, 72 (Study 105)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Arm 6: Part B LUM 400 mg q12h/ IVA 250 mg q12h | Arm 7: Part B Placebo- LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 55 | 60
kg
  Absolute Change at Day 15 | -0.1 (1.5) | -0.1 (1.8)
  Absolute Change at Week 8: number analyzed (Participants) | 54 | 57
  Absolute Change at Week 8 | 0 (2.3) | 0.4 (2.3)
  Absolute Change at Week 16: number analyzed (Participants) | 51 | 53
  Absolute Change at Week 16 | 0.3 (2.8) | 0.6 (2.9)
  Absolute Change at Week 24: number analyzed (Participants) | 39 | 37
  Absolute Change at Week 24 | 0.2 (2.6) | 0.4 (3)
  Absolute Change at Week 36: number analyzed (Participants) | 20 | 20
  Absolute Change at Week 36 | 0.3 (1.7) | 2.3 (3.3)
  Absolute Change at Week 48: number analyzed (Participants) | 17 | 17
  Absolute Change at Week 48 | 0.2 (2) | 2.2 (4.3)
  Absolute Change at Week 60: number analyzed (Participants) | 12 | 16
  Absolute Change at Week 60 | 0.3 (2.3) | 1.5 (3.3)
  Absolute Change at Week 72: number analyzed (Participants) | 13 | 15
  Absolute Change at Week 72 | 0.2 (2.3) | 1.1 (3.4)

15. Secondary Outcome: Part A Treatment Cohort: Time-to-First Pulmonary Exacerbation
Description: Time-to-first pulmonary exacerbation was analyzed using the Kaplan-Meier estimates. Pulmonary exacerbation was defined as the treatment with new or changed antibiotic therapy (intravenous, inhaled, or oral) for greater than or equal to 4 sinopulmonary signs/symptoms. Analysis was performed for the Cumulative Study Period for Arm 1 and 3, and for the current study period (Study 105) for Arm 2 and 4. As per planned analysis, endpoint evaluation included subjects from the parent study VX12-809-103 and VX12-809-104 as well for cumulative study period.
Time Frame: Baseline (Study 103/104) up to Week 100 (Study 105) for Arm 1 and 3 (Cumulative study period); Baseline (Study 105) up to Week 100 (Study 105) for Arm 2 and 4 (current study period)
Population: FAS (Study 103/104) was used for Arm 1 and 3, and included all participants randomized in the previous studies and dosed. FAS (Study 105) was used for Arm 2 and 4, and included all participants randomized in the Part A Treatment Cohort and dosed in current study 105.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Arm 1: Part A - LUM 600 mg qd/ IVA 250 mg q12h | Arm 2: Part A - Placebo- LUM 600 mg qd/ IVA 250 mg q12h | Arm 3: Part A - LUM 400 mg q12h/ IVA 250 mg q12h | Arm 4: Part A - Placebo- LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 368 | 179 | 369 | 176
days | 364 [99 to NA] — Data for Q3 interquartile range could not be estimated due to limited number of events. | 505 [111 to NA] — Data for Q3 interquartile range could not be estimated due to limited number of events. | 481 [132 to NA] — Data for Q3 interquartile range could not be estimated due to limited number of events. | 466 [153 to NA] — Data for Q3 interquartile range could not be estimated due to limited number of events.

16. Secondary Outcome: Part A Treatment Cohort: Percentage of Participants With at Least 1 Pulmonary Exacerbation
Description: Pulmonary exacerbation was defined as the treatment with new or changed antibiotic therapy (intravenous, inhaled, or oral) for greater than or equal to 4 sinopulmonary signs/symptoms. Analysis was performed for the Cumulative Study Period for Arm 1 and 3, and for the current study period (Study 105) for Arm 2 and 4. As per planned analysis, endpoint evaluation included subjects from the parent study VX12-809-103 and VX12-809-104 as well for cumulative study period.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: Part A - LUM 600 mg qd/ IVA 250 mg q12h | Arm 2: Part A - Placebo- LUM 600 mg qd/ IVA 250 mg q12h | Arm 3: Part A - LUM 400 mg q12h/ IVA 250 mg q12h | Arm 4: Part A - Placebo- LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 368 | 179 | 369 | 176
percentage of participants | 64.7 [59.8 to 69.6] | 53.6 [46.3 to 60.9] | 59.9 [54.9 to 64.9] | 55.7 [48.3 to 63]

17. Secondary Outcome: Part A Treatment Cohort: Percentage of Participants With Response Based on Relative Change in Percent Predicted FEV1 From Baseline
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Hankinson and Wang standards were used to calculate percent predicted FEV1 (for age, gender, race, and height). Percentage of participants with at least 5% and 10% relative change in percent predicted FEV1 from baseline were reported. Analysis was performed using baseline of the previous study VX12-809-103 (NCT01807923) and Study VX12-809-104 (NCT01807949) for Arm 1 and 3. Analysis was performed using baseline of the current study VX12-809-105 (NCT01931839) for Arm 2 and 4. As per planned analysis, endpoint evaluation included subjects from the parent study VX12-809-103 and VX12-809-104 as well for cumulative study period.
Time Frame: Baseline (Study 103/104/105); Day 15, Week 8, 16, 24, 36, 48, 60, 72, 84, 96 (Study 105)
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: Part A - LUM 600 mg qd/ IVA 250 mg q12h | Arm 2: Part A - Placebo- LUM 600 mg qd/ IVA 250 mg q12h | Arm 3: Part A - LUM 400 mg q12h/ IVA 250 mg q12h | Arm 4: Part A - Placebo- LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 368 | 179 | 369 | 176
percentage of participants
  Day 15: >=5% Change | 39.4 [34.4 to 44.4] | 42.5 [35.2 to 49.7] | 40.9 [35.9 to 45.9] | 42.6 [35.3 to 49.9]
  Day 15: >=10% Change | 25 [20.6 to 29.4] | 26.8 [20.3 to 33.3] | 24.7 [20.3 to 29.1] | 26.7 [20.2 to 33.2]
  Week 8: >=5% Change | 39.7 [34.7 to 44.7] | 38 [30.9 to 45.1] | 39.3 [34.3 to 44.3] | 48.9 [41.5 to 56.2]
  Week 8: >=10% Change | 26.9 [22.4 to 31.4] | 23.5 [17.3 to 29.7] | 26.6 [22.1 to 31.1] | 35.8 [28.7 to 42.9]
  Week 16: >=5% Change | 37.2 [32.3 to 42.2] | 36.9 [29.8 to 43.9] | 36.9 [31.9 to 41.8] | 46.6 [39.2 to 54]
  Week 16: >=10% Change | 25.5 [21.1 to 30] | 25.1 [18.8 to 31.5] | 26.3 [21.8 to 30.8] | 28.4 [21.7 to 35.1]
  Week 24: >=5% Change | 35.6 [30.7 to 40.5] | 38 [30.9 to 45.1] | 33.6 [28.8 to 38.4] | 42.6 [35.3 to 49.9]
  Week 24: >=10% Change | 24.5 [20.1 to 28.8] | 21.8 [15.7 to 27.8] | 22.5 [18.2 to 26.8] | 32.4 [25.5 to 39.3]
  Week 36: >=5% Change | 35.3 [30.4 to 40.2] | 32.4 [25.5 to 39.3] | 31.7 [27 to 36.5] | 38.6 [31.4 to 45.8]
  Week 36: >=10% Change | 23.4 [19 to 27.7] | 22.9 [16.7 to 29.1] | 22.2 [18 to 26.5] | 27.3 [20.7 to 33.9]
  Week 48: >=5% Change | 30.2 [25.5 to 34.9] | 32.4 [25.5 to 39.3] | 30.9 [26.2 to 35.6] | 36.4 [29.3 to 43.5]
  Week 48: >=10% Change | 21.7 [17.5 to 26] | 21.8 [15.7 to 27.8] | 21.4 [17.2 to 25.6] | 19.9 [14 to 25.8]
  Week 60: >=5% Change | 30.4 [25.7 to 35.1] | 32.4 [25.5 to 39.3] | 29.3 [24.6 to 33.9] | 38.6 [31.4 to 45.8]
  Week 60: >=10% Change | 20.4 [16.3 to 24.5] | 25.1 [18.8 to 31.5] | 19.2 [15.2 to 23.3] | 24.4 [18.1 to 30.8]
  Week 72: >=5% Change | 29.3 [24.7 to 34] | 34.6 [27.7 to 41.6] | 25.5 [21 to 29.9] | 33 [26 to 39.9]
  Week 72: >=10% Change | 18.2 [14.3 to 22.1] | 22.3 [16.2 to 28.4] | 18.2 [14.2 to 22.1] | 23.3 [17.1 to 29.5]
  Week 84: >=5% Change | 23.1 [18.8 to 27.4] | 28.5 [21.9 to 35.1] | 23.3 [19 to 27.6] | 26.1 [19.6 to 32.6]
  Week 84: >=10% Change | 14.9 [11.3 to 18.6] | 21.2 [15.2 to 27.2] | 15.7 [12 to 19.4] | 19.9 [14 to 25.8]
  Week 96: >=5% Change | 15.5 [11.8 to 19.2] | 14.5 [9.4 to 19.7] | 13.8 [10.3 to 17.3] | 15.3 [10 to 20.7]
  Week 96: >=10% Change | 8.7 [5.8 to 11.6] | 10.1 [5.7 to 14.5] | 10.3 [7.2 to 13.4] | 9.1 [4.8 to 13.3]

18. Secondary Outcome: Part B Treatment Cohort: Percentage of Participants With Response Based on Relative Change in Percent Predicted FEV1 From Baseline
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Hankinson and Wang standards were used to calculate percent predicted FEV1 (for age, gender, race, and height). Percentage of participants with at least 5% relative change in percent predicted FEV1 from Baseline were reported. Analysis was performed using baseline of Cohort 4 of previous study VX09-809-102 (NCT01225211) for Arm 6 and 7. As per planned analysis, endpoint evaluation included subjects from the parent study VX09-809-102 as well.
Time Frame: Baseline (Study 102), Day 15, Week 8, 16, 24, 36, 48, 60, 72 (Study 105)
Population: FAS (Study 102) was used for Arm 6 and 7, and included all participants randomized in the cohort 4 of study 102 and dosed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Arm 6: Part B LUM 400 mg q12h/ IVA 250 mg q12h: Participants who were randomized to LUM 400 mg plus IVA 250 mg FDC tablet orally in the morning and evening in Cohort 4 of the previous study VX09-809-102 (NCT01225211).
- Arm 7: Part B Placebo- LUM 400 mg q12h/ IVA 250 mg q12h: Participants who were randomized to placebo matched to LUM and IVA tablet in Cohort 4 of the previous study VX09-809-102 (NCT01225211).
Arm/Group | Arm 6: Part B LUM 400 mg q12h/ IVA 250 mg q12h | Arm 7: Part B Placebo- LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 62 | 63
percentage of participants
  Day 15: >=5% Change | 21 [10.8 to 31.1] | 12.7 [4.5 to 20.9]
  Week 8: >=5% Change | 11.3 [3.4 to 19.2] | 19 [9.4 to 28.7]
  Week 16: >=5% Change | 19.4 [9.5 to 29.2] | 15.9 [6.8 to 24.9]
  Week 24: >=5% Change | 12.9 [4.6 to 21.2] | 12.7 [4.5 to 20.9]
  Week 36: >=5% Change | 6.5 [0.3 to 12.6] | 6.3 [0.3 to 12.4]
  Week 48: >=5% Change | 6.5 [0.3 to 12.6] | 4.8 [0 to 10]
  Week 60: >=5% Change | 6.5 [0.3 to 12.6] | 6.3 [0.3 to 12.4]
  Week 72: >=5% Change | 3.2 [0 to 7.6] | 0 [0 to 0]
  Week 84: >=5% Change | 1.6 [0 to 4.7] | 1.6 [0 to 4.7]
  Week 96: >=5% Change | 0 [0 to 0] | 0 [0 to 0]

19. Secondary Outcome: Part A Observation Cohort: Number of Participants With Serious Adverse Events (SAEs)
Description: AE: as any untoward medical occurrence in a participant during the study; the event does not necessarily have a causal relationship with the treatment. This includes any newly occurring event or previous condition that has increased in severity or frequency after the informed consent form is signed. AE includes serious as well as non-serious AEs. SAE (subset of AE): medical event or condition, which falls into any of the following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, In-patient hospitalization/prolongation of hospitalization, persistent/significant disability or incapacity, congenital anomaly/birth defect, important medical event.
Time Frame: up to 2 years
Population: Safety Set (study 105) included all participants who were enrolled in Part A Observation Cohort.
Measure: Number; unit: participants
Groups:
- Arm 5: Part A Observational Cohort: Participants who received either LUM 600 mg plus IVA 250 mg FDC tablet orally in the morning and IVA 250 mg film-coated tablet orally in the evening or LUM 400 mg plus IVA 250 mg FDC tablet orally in the morning and evening or placebo matched to LUM and IVA in the morning and evening, in the previous study VX12-809-103 (NCT01807923) or VX12-809-104 (NCT01807949), were observed (did not receive study drug) in this study VX12-809-105 (NCT01931839) for up to 2 years.
Arm/Group | Arm 5: Part A Observational Cohort
Number analyzed (Participants) | 19
participants | 7

ADVERSE EVENTS:
Description: Non-SAEs were not collected for Arm 5: Part A Observational Cohort. Only SAEs were collected.
Arm/Group | Arm 1 Part A: LUM 600 mg qd/ IVA 250 mg q12h | Arm 2 Part A: Placebo - LUM 600 mg qd/ IVA 250 mg q12h | Arm 3 Part A: LUM 400 mg q12h/ IVA 250 mg q12h | Arm 4 Part A: Placebo - LUM 400 mg q12h/ IVA 250 mg q12h | Arm 5 Part A: Observational Cohort | Arm 6 Part B: LUM 400 mg q12h/ IVA 250 mg q12h | Arm 7 Part B: Placebo - LUM 400 mg q12h/ IVA 250 mg q12h
Serious Adverse Events (participants affected / at risk) | 156/335 | 77/178 | 143/340 | 89/176 | 7/19 | 18/55 | 21/60
Other Adverse Events (participants affected / at risk) | 328/335 | 177/178 | 332/340 | 173/176 | 0/0 | 52/55 | 57/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 Part A: LUM 600 mg qd/ IVA 250 mg q12h (N=335) | Arm 2 Part A: Placebo - LUM 600 mg qd/ IVA 250 mg q12h (N=178) | Arm 3 Part A: LUM 400 mg q12h/ IVA 250 mg q12h (N=340) | Arm 4 Part A: Placebo - LUM 400 mg q12h/ IVA 250 mg q12h (N=176) | Arm 5 Part A: Observational Cohort (N=19) | Arm 6 Part B: LUM 400 mg q12h/ IVA 250 mg q12h (N=55) | Arm 7 Part B: Placebo - LUM 400 mg q12h/ IVA 250 mg q12h (N=60)
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Serum sickness (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Type IV hypersensitivity reaction (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Medical device site thrombosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary function test decreased (Investigations) | 3 | 1 | 3 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 2 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 2 | 0 | 0 | 0
Bacterial test positive (Investigations) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Forced expiratory volume decreased (Investigations) | 0 | 0 | 0 | 3 | 0 | 1 | 0
Gammaglutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza B virus test positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza A virus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cystic fibrosis related diabetes (Congenital, familial and genetic disorders) | 2 | 0 | 3 | 3 | 0 | 0 | 1
Cystic fibrosis pancreatic (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 17 | 7 | 10 | 6 | 1 | 0 | 2
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 3 | 0 | 0 | 0 | 0
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 3 | 0 | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary bulla (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cauda equina syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Juvenile myoclonic epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neurological symptom (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vocal cord paralysis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cataract subcapsular (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 2 | 1 | 6 | 10 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 5 | 1 | 1 | 2 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mechanical ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 113 | 61 | 111 | 59 | 5 | 15 | 15
Pneumonia (Infections and infestations) | 6 | 4 | 5 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 2 | 6 | 3 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 3 | 2 | 1 | 1 | 0 | 0 | 0
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Device related sepsis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 1
Respiratory tract infection bacterial (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Tracheobronchitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatitis E (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung infection pseudomonal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mediastinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mycobacterium abscessus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Parotitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Periorbital abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 Part A: LUM 600 mg qd/ IVA 250 mg q12h (N=335) | Arm 2 Part A: Placebo - LUM 600 mg qd/ IVA 250 mg q12h (N=178) | Arm 3 Part A: LUM 400 mg q12h/ IVA 250 mg q12h (N=340) | Arm 4 Part A: Placebo - LUM 400 mg q12h/ IVA 250 mg q12h (N=176) | Arm 5 Part A: Observational Cohort (N=0) | Arm 6 Part B: LUM 400 mg q12h/ IVA 250 mg q12h (N=55) | Arm 7 Part B: Placebo - LUM 400 mg q12h/ IVA 250 mg q12h (N=60)
Contusion (Injury, poisoning and procedural complications) | 7 | 3 | 8 | 3 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 10 | 3 | 8 | 0 | 0 | 0 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 5 | 2 | 5 | 6 | 0 | 2 | 0
Muscle strain (Injury, poisoning and procedural complications) | 5 | 4 | 2 | 1 | 0 | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 4 | 3 | 3 | 1 | 0 | 2 | 0
Laceration (Injury, poisoning and procedural complications) | 2 | 3 | 5 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 5 | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 2 | 1 | 3 | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 3 | 0 | 4 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 4 | 0 | 2 | 1 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 1 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 2 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 4 | 0 | 2 | 0 | 0 | 1 | 0
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 2 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 5 | 0 | 0 | 1 | 0 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 3 | 0 | 2 | 0 | 0 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 1 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 2 | 0 | 0 | 0
Back injury (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Sports injury (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Superficial injury of eye (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Stoma site discomfort (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Stoma site irritation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Animal scratch (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Confusion postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Heat stroke (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Incision site haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lip injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neck injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nerve injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral nerve injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Procedural anxiety (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Procedural headache (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus barotrauma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Splinter (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stoma site erythema (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stoma site pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stoma site ulcer (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stress fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary function test decreased (Investigations) | 35 | 23 | 29 | 15 | 0 | 2 | 3
Blood creatine phosphokinase increased (Investigations) | 26 | 23 | 23 | 15 | 0 | 5 | 10
Forced expiratory volume decreased (Investigations) | 26 | 12 | 28 | 15 | 0 | 2 | 7
Bacterial test positive (Investigations) | 29 | 7 | 30 | 11 | 0 | 2 | 1
Alanine aminotransferase increased (Investigations) | 10 | 14 | 14 | 15 | 0 | 2 | 4
Aspartate aminotransferase increased (Investigations) | 12 | 13 | 15 | 13 | 0 | 1 | 7
Blood glucose decreased (Investigations) | 4 | 1 | 4 | 2 | 0 | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 1 | 3 | 2 | 0 | 1 | 1
Weight decreased (Investigations) | 16 | 7 | 18 | 3 | 0 | 2 | 0
Blood creatinine increased (Investigations) | 5 | 6 | 3 | 7 | 0 | 1 | 1
Blood glucose increased (Investigations) | 5 | 7 | 2 | 6 | 0 | 0 | 1
Fungal test positive (Investigations) | 5 | 4 | 6 | 2 | 0 | 1 | 0
Vitamin D decreased (Investigations) | 6 | 3 | 3 | 5 | 0 | 0 | 0
Liver function test increased (Investigations) | 1 | 6 | 3 | 2 | 0 | 0 | 1
White blood cell count increased (Investigations) | 4 | 5 | 2 | 1 | 0 | 0 | 1
Atypical mycobacterium test positive (Investigations) | 3 | 5 | 2 | 1 | 0 | 0 | 0
Influenza A virus test positive (Investigations) | 3 | 3 | 3 | 2 | 0 | 1 | 0
Neutrophil count increased (Investigations) | 2 | 3 | 3 | 1 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 3 | 1 | 3 | 0 | 0 | 0 | 2
Blood magnesium decreased (Investigations) | 2 | 2 | 1 | 0 | 0 | 0 | 0
Clostridium test positive (Investigations) | 2 | 1 | 1 | 1 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 2 | 0 | 2 | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 2 | 2 | 1 | 0 | 0 | 0 | 0
White blood cells urine positive (Investigations) | 2 | 0 | 2 | 1 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 2 | 1 | 0 | 0 | 1 | 0
Blood bicarbonate decreased (Investigations) | 2 | 1 | 0 | 1 | 0 | 0 | 0
Blood immunoglobulin E increased (Investigations) | 1 | 1 | 1 | 1 | 0 | 0 | 0
Body temperature increased (Investigations) | 1 | 0 | 1 | 2 | 0 | 0 | 0
Crystal urine present (Investigations) | 2 | 0 | 1 | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 2 | 0 | 1 | 1 | 0 | 0 | 0
Protein urine present (Investigations) | 0 | 0 | 2 | 2 | 0 | 0 | 0
Staphylococcus test positive (Investigations) | 1 | 1 | 1 | 1 | 0 | 0 | 0
Blood calcium increased (Investigations) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 1 | 2 | 0 | 0 | 0
Blood pressure systolic increased (Investigations) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 1 | 2 | 0 | 0 | 0
Forced vital capacity decreased (Investigations) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Glucose urine present (Investigations) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Monocyte count increased (Investigations) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Pseudomonas test positive (Investigations) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Candida test positive (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Glucose tolerance test abnormal (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Human rhinovirus test positive (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Influenza B virus test positive (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood immunoglobulin G increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood iron decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Helicobacter test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza virus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 1
Reticulocyte percentage increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sputum abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Platelet count increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory syncytial virus test positive (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Aspergillus test positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood androstenedione increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood cortisol decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood glucose fluctuation (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood magnesium increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood phosphorus increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood sodium decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood sodium increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood testosterone decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood testosterone increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood urine present (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Burkholderia test positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Citrobacter test positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Computerised tomogram thorax abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Coronavirus test positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydroepiandrosterone increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram PR shortened (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram ST segment elevation (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epstein-Barr virus antibody positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Escherichia test positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Grip strength decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemoglobin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Human metapneumovirus test positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Human papilloma virus test positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mean cell volume increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myoglobin blood increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Precancerous cells present (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Red blood cells urine positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Reticulocyte count increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rubulavirus test positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ultrasound liver abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urine analysis abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urine bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urine ketone body present (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral test positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitamin A decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vitamin B12 decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitamin E decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cyanosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 5 | 0 | 4 | 2 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 1 | 3 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thyroglossal cyst (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystic fibrosis related diabetes (Congenital, familial and genetic disorders) | 10 | 10 | 8 | 5 | 0 | 0 | 0
Cystic fibrosis hepatic disease (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cystic fibrosis lung (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Naevus flammeus (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 7 | 1 | 5 | 2 | 0 | 1 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 1 | 0 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Bone marrow oedema (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemoconcentration (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Macrocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 58 | 25 | 56 | 22 | 0 | 7 | 7
Sinus headache (Nervous system disorders) | 13 | 9 | 11 | 3 | 0 | 2 | 2
Dizziness (Nervous system disorders) | 9 | 7 | 6 | 6 | 0 | 1 | 1
Migraine (Nervous system disorders) | 6 | 2 | 5 | 2 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 2 | 1 | 2 | 4 | 0 | 0 | 0
Syncope (Nervous system disorders) | 2 | 1 | 2 | 2 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 3 | 0 | 3 | 2 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 4 | 0 | 3 | 0 | 0 | 0 | 0
Anosmia (Nervous system disorders) | 3 | 0 | 0 | 2 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0
Circadian rhythm sleep disorder (Nervous system disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Migraine with aura (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aphonia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coordination abnormal (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyposmia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intercostal neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Olfactory nerve disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1
Blepharospasm (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1
Conjunctivitis allergic (Eye disorders) | 2 | 2 | 4 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 5 | 0 | 0 | 0
Dry eye (Nervous system disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0
Eye pruritus (Nervous system disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0
Lacrimation increased (Nervous system disorders) | 1 | 0 | 3 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Diabetic retinopathy (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myopia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ulcerative keratitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 6 | 6 | 5 | 4 | 0 | 0 | 2
Tinnitus (Ear and labyrinth disorders) | 5 | 6 | 1 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 2 | 3 | 2 | 0 | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear pruritus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Middle ear effusion (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Motion sickness (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ototoxicity (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 46 | 24 | 41 | 28 | 0 | 5 | 9
Nausea (Gastrointestinal disorders) | 45 | 24 | 34 | 27 | 0 | 5 | 4
Abdominal pain (Gastrointestinal disorders) | 42 | 20 | 33 | 15 | 0 | 3 | 2
Constipation (Gastrointestinal disorders) | 28 | 13 | 24 | 10 | 0 | 3 | 3
Vomiting (Gastrointestinal disorders) | 26 | 6 | 27 | 13 | 0 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 18 | 9 | 20 | 11 | 0 | 6 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 16 | 8 | 14 | 4 | 0 | 5 | 2
Flatulence (Gastrointestinal disorders) | 13 | 5 | 7 | 7 | 0 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 8 | 5 | 10 | 6 | 0 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 11 | 2 | 10 | 4 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 3 | 4 | 7 | 3 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 4 | 1 | 5 | 4 | 0 | 0 | 1
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 3 | 5 | 5 | 1 | 0 | 0 | 0
Dental discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post-tussive vomiting (Gastrointestinal disorders) | 1 | 3 | 1 | 2 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 3 | 3 | 4 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 3 | 3 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 1 | 4 | 0 | 0 | 0 | 0
Steatorrhoea (Gastrointestinal disorders) | 2 | 0 | 2 | 2 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 2 | 1 | 1 | 2 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Tooth impacted (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Bowel movement irregularity (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Breath odour (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Faecal volume decreased (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Faecal volume increased (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastric mucosal hypertrophy (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gingival erythema (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gingival recession (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Glossitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intussusception (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malabsorption (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malpositioned teeth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mucous stools (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oesophageal irritation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oesophageal mucosal hyperplasia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oesophageal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral papule (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatic insufficiency (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Reflux gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth delamination (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 3 | 3 | 2 | 2 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Glycosuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypernatriuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypocitraturia (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyelocaliectasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal hypertrophy (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal pain (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal tubular disorder (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urine abnormality (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 10 | 9 | 22 | 7 | 0 | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 3 | 3 | 8 | 7 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 3 | 6 | 6 | 0 | 0 | 4
Night sweats (Skin and subcutaneous tissue disorders) | 5 | 7 | 4 | 2 | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 6 | 5 | 5 | 2 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 3 | 3 | 4 | 0 | 2 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 4 | 6 | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 5 | 1 | 4 | 0 | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 5 | 3 | 1 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 2 | 3 | 1 | 0 | 0 | 0
Red man syndrome (Skin and subcutaneous tissue disorders) | 1 | 3 | 3 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 2 | 0 | 0 | 0
Pruritus allergic (Skin and subcutaneous tissue disorders) | 4 | 0 | 1 | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 4 | 1 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 5 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 1 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 2 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 0 | 1 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Skin warm (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Solar dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Acne cystic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fixed drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Madarosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Purpura senile (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash morbilliform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Scar pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin wrinkling (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urticarial vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Device dislocation (Product Issues) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Device occlusion (Product Issues) | 4 | 1 | 2 | 0 | 0 | 0 | 0
Device leakage (Product Issues) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 | 11 | 25 | 13 | 0 | 3 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 12 | 14 | 10 | 0 | 1 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 19 | 7 | 13 | 5 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 13 | 9 | 12 | 3 | 0 | 2 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 | 6 | 5 | 6 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 5 | 7 | 2 | 0 | 2 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 2 | 7 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 1 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 1 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 4 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 | 0 | 0 | 2 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 0 | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc annular tear (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mastication disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle oedema (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Growth hormone deficiency (Endocrine disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Androgen deficiency (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cushing's syndrome (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 11 | 5 | 16 | 6 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 12 | 8 | 6 | 9 | 0 | 2 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 7 | 3 | 3 | 0 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 4 | 3 | 0 | 0 | 1 | 3
Iron deficiency (Metabolism and nutrition disorders) | 6 | 1 | 3 | 2 | 0 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 3 | 1 | 2 | 2 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 3 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 | 0 | 1 | 1
Alcohol intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3 | 1 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypovitaminosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Selenium deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vitamin A deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Vitamin E deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 2 | 1 | 2 | 1 | 0 | 0 | 0
Vitamin K deficiency (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyponatraemic syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Underweight (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight gain poor (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 185 | 92 | 173 | 91 | 0 | 18 | 20
Nasopharyngitis (Infections and infestations) | 51 | 31 | 66 | 27 | 0 | 6 | 6
Upper respiratory tract infection (Infections and infestations) | 42 | 26 | 49 | 29 | 0 | 7 | 6
Sinusitis (Infections and infestations) | 41 | 19 | 47 | 13 | 0 | 7 | 2
Viral upper respiratory tract infection (Infections and infestations) | 34 | 12 | 24 | 10 | 0 | 3 | 4
Influenza (Infections and infestations) | 20 | 11 | 21 | 15 | 0 | 2 | 1
Rhinitis (Infections and infestations) | 24 | 7 | 21 | 12 | 0 | 1 | 1
Upper respiratory tract infection bacterial (Infections and infestations) | 16 | 14 | 18 | 7 | 0 | 2 | 1
Bronchitis (Infections and infestations) | 15 | 8 | 12 | 8 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 21 | 4 | 7 | 9 | 0 | 1 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 13 | 4 | 14 | 7 | 0 | 2 | 2
Respiratory tract infection viral (Infections and infestations) | 11 | 4 | 11 | 3 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 10 | 3 | 5 | 8 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 8 | 6 | 7 | 5 | 0 | 2 | 0
Respiratory tract infection (Infections and infestations) | 6 | 6 | 7 | 6 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 8 | 2 | 7 | 5 | 0 | 2 | 1
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 9 | 6 | 4 | 2 | 0 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 4 | 4 | 6 | 6 | 0 | 2 | 1
Otitis media (Infections and infestations) | 9 | 1 | 8 | 1 | 0 | 2 | 0
Gastroenteritis viral (Infections and infestations) | 12 | 2 | 4 | 0 | 0 | 1 | 0
Lung infection pseudomonal (Infections and infestations) | 5 | 3 | 6 | 3 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 5 | 1 | 5 | 4 | 0 | 2 | 1
Chronic sinusitis (Infections and infestations) | 4 | 4 | 5 | 1 | 0 | 1 | 0
Respiratory tract infection bacterial (Infections and infestations) | 9 | 2 | 2 | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 5 | 1 | 5 | 3 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 6 | 1 | 2 | 4 | 0 | 0 | 0
Viral infection (Infections and infestations) | 5 | 2 | 5 | 1 | 0 | 1 | 1
Pharyngitis streptococcal (Infections and infestations) | 7 | 1 | 4 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 3 | 1 | 5 | 2 | 0 | 0 | 3
Bacterial disease carrier (Infections and infestations) | 3 | 0 | 5 | 2 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 4 | 2 | 2 | 2 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 4 | 3 | 1 | 0 | 0 | 0
Lower respiratory tract infection bacterial (Infections and infestations) | 4 | 1 | 3 | 1 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 2 | 3 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 4 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 2 | 1 | 3 | 1 | 0 | 0 | 0
Lower respiratory tract infection viral (Infections and infestations) | 3 | 2 | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 2 | 0 | 2 | 2 | 0 | 0 | 3
Folliculitis (Infections and infestations) | 2 | 0 | 2 | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 4 | 0 | 0 | 0 | 0
Bronchitis viral (Infections and infestations) | 1 | 2 | 0 | 1 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 2 | 0 | 1 | 1 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 2 | 0 | 1 | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 3 | 1 | 0 | 0 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Eye infection (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Genital candidiasis (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Herpes dermatitis (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Sinusitis bacterial (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Stoma site infection (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Tinea infection (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Bronchitis bacterial (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Infectious mononucleosis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Mycobacterial disease carrier (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Superinfection bacterial (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Mycobacterium abscessus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngitis fungal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Otitis externa fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Parotitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 1 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Viral pharyngitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acne pustular (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Adenoiditis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Angular cheilitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atypical mycobacterial lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atypical mycobacterial pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis fungal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epididymitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erythema infectiosum (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Febrile infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Genital herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Genital herpes simplex (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Genital infection fungal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Groin abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemophilus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Helicobacter infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis C (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Implant site infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Labyrinthitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Overgrowth bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Overgrowth fungal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Papilloma viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pseudomonas bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulpitis dental (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Salpingo-oophoritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection fungal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Small intestinal bacterial overgrowth (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sputum purulent (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Trichomoniasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory fungal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 3 | 2 | 4 | 3 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 1 | 2 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Vasodilatation (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ethmoid sinus surgery (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wisdom teeth removal (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neurofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 13 | 5 | 19 | 5 | 0 | 3 | 3
Drug hypersensitivity (Immune system disorders) | 4 | 3 | 4 | 4 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0
Allergy to arthropod bite (Immune system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Allergy to animal (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
House dust allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Immunisation reaction (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mycotic allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Reaction to food additive (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Serum sickness (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Smoke sensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Menopause (Social circumstances) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 60 | 27 | 47 | 31 | 0 | 6 | 8
Fatigue (General disorders) | 45 | 26 | 36 | 22 | 0 | 7 | 6
Pain (General disorders) | 12 | 5 | 6 | 3 | 0 | 1 | 1
Malaise (General disorders) | 3 | 4 | 9 | 1 | 0 | 1 | 1
Chest discomfort (General disorders) | 7 | 6 | 3 | 7 | 0 | 0 | 0
Chest pain (General disorders) | 7 | 6 | 2 | 4 | 0 | 0 | 1
Asthenia (General disorders) | 6 | 2 | 5 | 2 | 0 | 0 | 1
Chills (General disorders) | 4 | 3 | 6 | 1 | 0 | 0 | 1
Influenza like illness (General disorders) | 2 | 2 | 5 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 3 | 1 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0
Feeling cold (General disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Application site vesicles (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Catheter site haematoma (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Exercise tolerance decreased (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 2
Sensation of foreign body (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Application site irritation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Catheter site rash (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug intolerance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug withdrawal syndrome (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Facial pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hernia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hunger (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion site bruising (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion site pruritus (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mass (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Medical device pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Medical device site ulcer (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Temperature intolerance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaccination site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site phlebitis (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infusion site inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Medical device site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 14 | 5 | 9 | 3 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 7 | 9 | 9 | 2 | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 0 | 3 | 2 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 4 | 1 | 0 | 0 | 0 | 0 | 0
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Stress (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Adjustment disorder (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Adjustment disorder with anxiety (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased interest (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Disturbance in social behaviour (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Encopresis (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Food aversion (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Listless (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Obsessive-compulsive disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Somnambulism (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 7 | 4 | 8 | 10 | 0 | 1 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 6 | 3 | 8 | 4 | 0 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 6 | 2 | 2 | 3 | 0 | 0 | 0
Abnormal withdrawal bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cervical polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 1 | 2 | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 3 | 1 | 3 | 2 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 1 | 1 | 2 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 3 | 0 | 0 | 0 | 0
Polycystic ovaries (Reproductive system and breast disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Acquired hydrocele (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Adnexa uteri mass (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Amenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bartholin's cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ovarian hyperfunction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Polymenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus genital (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectocele (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Testicular cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 167 | 92 | 145 | 82 | 0 | 18 | 18
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 75 | 36 | 79 | 37 | 0 | 11 | 18
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 61 | 37 | 68 | 29 | 0 | 8 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 52 | 33 | 53 | 36 | 0 | 9 | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 45 | 21 | 44 | 22 | 0 | 8 | 7
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 39 | 30 | 34 | 25 | 0 | 7 | 21
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 40 | 20 | 37 | 23 | 0 | 8 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 20 | 10 | 21 | 13 | 0 | 2 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 22 | 9 | 18 | 12 | 0 | 7 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 26 | 8 | 12 | 7 | 0 | 2 | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 16 | 7 | 13 | 12 | 0 | 3 | 3
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 14 | 4 | 18 | 7 | 0 | 3 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 19 | 5 | 14 | 3 | 0 | 5 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 13 | 6 | 16 | 5 | 0 | 2 | 1
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 20 | 3 | 12 | 5 | 0 | 0 | 4
Rales (Respiratory, thoracic and mediastinal disorders) | 10 | 9 | 10 | 11 | 0 | 1 | 2
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 13 | 4 | 12 | 6 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 9 | 2 | 12 | 7 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 10 | 2 | 10 | 6 | 0 | 0 | 3
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 8 | 8 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 9 | 10 | 7 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 2 | 10 | 4 | 0 | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 8 | 9 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 10 | 5 | 4 | 6 | 0 | 1 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 6 | 4 | 0 | 1 | 1
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 4 | 2 | 0 | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 5 | 2 | 0 | 1 | 0
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 3 | 1 | 0 | 0 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 5 | 1 | 0 | 1 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 5 | 0 | 0 | 0 | 0
Nasal discharge discolouration (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 4 | 1 | 0 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 0 | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0 | 0 | 0 | 0 | 2
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3 | 1 | 0 | 1 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 0 | 0 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 5 | 0 | 0 | 0
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 0 | 0 | 0 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 0 | 0 | 0 | 0
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 0 | 0 | 0 | 0
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Acquired diaphragmatic eventration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Allergic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchial irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Increased viscosity of upper respiratory secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung hyperinflation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary bulla (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tonsillolith (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tracheal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tracheal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Analysis using baseline values of the current study 105 (NCT01931839) was not performed for Part B Treatment Cohort.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is free to publish results of the study after (1) the first multi-center publication, (2) if the sponsor elects not to publish the results, or (3) 18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.